CLINICAL TRIAL: NCT01318564
Title: Treatment Adherence With Compliance Prompting Packaging
Brief Title: Diabetic Treatment Adherence
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2008-0242; U18HS016093 (AHRQ)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Endocrine System Diseases
Keywords: Type II Diabetes; Unit dose packaging devices; Metformin; Lisinopril; Enalapril; Atorvastatin; Lipitor; Simvastatin; Aspirin; Questionnaires
MeSH Terms: conditions — Endocrine System Diseases; Diabetes Mellitus, Type 2 | interventions — Metformin; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A fasting blood sample of 10 ml will be collected 2 days after randomization if the physician considers the test as a standard of care.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Unit-dose - Pill Bottle: Unit-dose (blister) packages used first week, followed second week by pill bottles usage.
  Interventions: Drug: Metformin; Behavioral: Questionnaires
- Group 2: Pill Bottle - Unit Dose: Pill bottle usage the first week followed second week by Unit-dose (blister) packages.
  Interventions: Drug: Metformin; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Metformin — 500 - 1000 mg by mouth twice a day with either via a MEMS device pill bottle (medication event monitoring system) or by unit-dosing (blister packaging) with attached Med-ic device (electronic compliance monitoring for blistered medication).
Behavioral: Questionnaires — Completion on Day 1 and after Month 3. Each questionnaire to take about 30 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to test an investigational type of packaging for diabetes drugs called "unit-dose packaging." Researchers want to learn if unit-dose packaging can help patients with Type II diabetes to take their drugs on the proper schedule.

DETAILED DESCRIPTION:
Study Background:

Some people find it difficult to take drugs on the proper schedule. For this reason, researchers want to learn if a different kind of drug packaging can help patients take their drugs more easily.

In unit-dose packaging, each pill is packaged in its own plastic bubble (called a "blister") on a package that has a calendar on it. This is designed to make it easier to keep track of when the pills should be taken.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will keep taking the same drugs that you are taking now. You will also keep taking those drugs on the same schedule that your doctor prescribed. The specific "study drugs" you may be taking are metformin, lisinopril, enalapril, atorvastatin, simvastatin, and aspirin.

You will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You have an equal chance of being assigned to either group.

Group 1 will receive their study drugs in unit-dose packages (also called "reminder blister packages") from Visit 1 to Visit 2.

Group 2 will receive their study drugs in pill bottles from Visit 1 to Visit 2.

Data Collection on Pill Usage:

There are electronic sensors on each blister package and pill bottle. If you are using blister packages (Group 1), the sensors will record the dates and times that you remove pills from the blisters. If you are using pill bottles (Group 2), the sensors will record the dates and times that you open the bottles.

It is important that you do not remove the pills too early before your dose (for example, the night before), so that the proper time is recorded.

You should return the empty blister packages or bottles to the clinic at each study visit. When you return the empty packaging, researchers will be able to collect the data that the sensors recorded (times and dates).

Study Visits:

On Day 1 and after Month 3, you will complete a questionnaire. It includes questions about your overall health, daily activities, and moods. There are also questions about how you take your drugs and how you feel about your diabetes drugs such as metformin. This questionnaire should take about 30-45 minutes to complete.

Researchers will record the results of your routine blood sugar level tests performed on Day 1 and after Month 3. Researchers will also record the results of your routine cholesterol level blood tests on Day 1 and after Month 3. The purpose is to learn how the drugs may impact your health status.

At each visit your blood pressure will be measured 3 times. This will take about 15 min. If your questionnaire responses show that you may be having emotional difficulties or depression, you will receive contact information for the counseling staff in case you would like to speak with a counselor.

Study Databases:

Your questionnaire and blood test data will be kept confidential and will only be used for this study. The same is true for the pill/package usage data recorded by the electronic sensors.

The study data will be entered into password-protected databases. In the databases, your name and other identifying information will not be used. Instead, your study identification (ID) number will be used.

Length of Study Participation:

Your study participation will be over after you complete the questionnaire after Month 3.

This is an investigational study. Unit-dose packaging is an FDA-approved type of packing for certain other drugs. At this time and for these particular drugs, unit-dose packaging is only being used in research.

Up to 120 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of 18 years or older.
2. Patients with type II Diabetes taking or eligible to start metformin with at least another medication for hypertension (Lisinopril or Enalapril), hyperlipidemia (atorvastatin or simvastatin) and/or aspirin.

Exclusion Criteria:

1. Dementia
2. Patients receiving current intravenous chemotherapy
3. Pregnancy
4. Patients residing in a nursing home
5. Treatment with any type of Insulin
6. Patients wanting to continue to use pill organizers for monitored medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Internal Medicine/Ambulatory Clinics at UT MD Anderson Cancer Center in Houston, Texas Kelsey-Seybold Outpatient Clinics in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Patients' Adherence to Unit Dose Packaging Devices | 12 weeks
  Taking information from the electronic monitor device packages, adherence considered as a ratio of prescribed doses to doses taken.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Suarez-Almazor, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Kelsey Seybold Clinics, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org